CLINICAL TRIAL: NCT00891631
Title: Primary Care Internet/Intranet-based Screening, Brief Intervention, and Referral to Treatment (iSBIRT) System to Reduce Serious Teen Health Risks
Brief Title: Primary Care iSBIRT to Reduce Serious Teen Health Risks
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Grant application was not funded
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, John R Knight, MD, Associate Professor of Pediatrics, Harvard Medical School; Senior Associate in Medicine; Associate in Psychiatry, Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: iSBIRT RFA-od-09-003
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Substance-related Disorders; Depression; High-risk Sex
Keywords: tobacco; alcohol; marijuana; drug use; seat-belt; weapons; depression; suicidality; sexual risk behaviors
MeSH Terms: conditions — Substance-Related Disorders; Depression; Unsafe Sex; Marijuana Abuse; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- iSBIRT (Experimental): Participants will complete the iSBIRT system.
  Interventions: Behavioral: iSBIRT
- iSBIRT/TE (Experimental): Participants will receive the internet/intranet screening, brief intervention, and referral to treatment system and technological extenders
  Interventions: Behavioral: iSBIRT/TE
- TAU (No Intervention): Participants will receive Treatment as Usual from their primary care provider.

INTERVENTIONS:
Behavioral: iSBIRT — Participants will receive the internet/intranet based screening, brief intervention, and referral to treatment program.
  Other Names: SBIRT
  Arms: iSBIRT
Behavioral: iSBIRT/TE — Participants will receive the internet/intranet screening, brief intervention, and referral to treatment system along with technological extenders
  Other Names: SBIRT
  Arms: iSBIRT/TE

SUMMARY:
The goal of the project is to develop and test an internet/intranet-based Screening, Brief Intervention, and Referral to Treatment (iSBIRT) system for adolescents that targets a broad range of serious health-risks and problem behaviors.

DETAILED DESCRIPTION:
We have previously developed and tested a computerized substance use screening and feedback program for adolescents. We will expand this program to include other serious health risks, enhance the feedback and health risk information adolescents will receive on the computer, develop Technological Extenders to extend the effect of the intervention, develop a training video and protocol for providers, and pilot test the system among adolescents coming for non-urgent care at a variety of primary care sites.

ELIGIBILITY:
Inclusion Criteria:

* 12-21 years old
* arriving for non-urgent care
* provide informed assent/consent

Exclusion Criteria:

* less than 6th grade reading level
* unavailable for follow-up questionnaires

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
frequency of substance use and other risk behaviors | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: John R Knight, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web site of the Center for Adolescent Substance Abuse Research at Children's Hospital Boston — http://www.ceasar.org